CLINICAL TRIAL: NCT03143023
Title: Efficacy of Dentifrices Containing Arginine Versus Fluoride on Microbial Acid Using Chair Side(Potential of Hydrogen) pH Meter Assessment Method in Adult Population: Randomized Clinical Trial
Brief Title: Efficacy of Dentifrices Containing Arginine Versus Fluoride on Microbial Acid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Laura Yehia, Resident of conservative departement , Faculty of Oral and Dental Medicine, Cairo university,2013, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBC-CU-2017-04-18
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arginine toothpaste (Experimental)
  Interventions: Drug: arginine toothpaste
- fluoride toothpaste (Active Comparator)
  Interventions: Drug: fluoride toothpaste

INTERVENTIONS:
Drug: arginine toothpaste — acid neutralizer toothpaste
  Arms: arginine toothpaste
Drug: fluoride toothpaste — bactericidal toothpaste
  Arms: fluoride toothpaste

SUMMARY:
This study will be conducted to evaluate the effect of arginine versus fluoride containing toothpaste on neutralization of microbial acid produced by Cariogenic bacteria in adult population using chair side assessment method.

DETAILED DESCRIPTION:
.28 volunteer participants will be assigned in this study. Participants will be randomly divided into two groups(n=14) according to type of toothpaste D where groups D1 patient will use arginine containing toothpaste while groups D2 the patient will used the fluoride toothpaste with a number of 14 patients in each group. The pH will be evaluated according to time in relation to the brushing with toothpaste (T) where (T0) represent salivary pH before brushing with toothpaste , (T1) represent salivary pH 10 minutes after brushing with toothpaste at fixed time of the day.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be over 18 years of age.
* Systematically healthy.
* Not taking any medication interfering with saliva secretion.
* Participants who signed informed consent.

Exclusion Criteria:

* Participants with a compromised medical history.
* Participants under systemic disease treatment, with antibiotic, steroid or any medication known to cause dry mouth.
* Severe or active periodontal disease.
* History of allergies or other adverse reactions to arginine, or oral care product or their ingredient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
salivary pH | 10 minutes after intervention and control
  Salivary pH will be determined by use of a digital pH meter .All salivary pH values will be taken immediately following salivary collection at chairside. The salivary pH values measured before usage of toothpaste termed "resting pH," while the salivary pH values measured after usage of toothpaste termed "terminal pH.

IPD SHARING:
Plan to Share IPD: Undecided